CLINICAL TRIAL: NCT01834807
Title: Retrospective Study on the Use of Biologicals in Monotherapy in Rheumatoid Arthritis
Brief Title: A Retrospective Observational Study on the Use of Biologics in Monotherapy in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28540
Record Dates: First submitted 2013-04-11; First posted 2013-04-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This retrospective, observational, multi-center study will evaluate the use of biological agents (e.g. RoActemra/Actemra [tocilizumab]) in monotherapy in patients with rheumatoid arthritis. Data from medical record files will be collected of patients currently treated with a biologic in monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Diagnosis of rheumatoid arthritis
* Currently receiving a biologic agent in monotherapy (corticosteroids and/or non-steroidal anti-inflammatory drugs are permitted)

Exclusion Criteria:

* Concomitant treatment with disease-modifying anti-rheumatic drugs (DMARDs) for the treatment of rheumatoid arthritis
* Patients that have started their current monotherapy before 01/01/2009

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis who are currently receiving a biologic agent in monotherapy (corticosteroids and/or non-steroidal anti-inflammatory drugs are permitted)
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Treatment schedule/duration of biological agents used in monotherapy in routine clinical practice | approximately 1 year
Type of biological agents used in monotherapy in routine clinical practice | approximately 1 year

SECONDARY OUTCOMES:
Efficacy: Response according to DAS28-ESR/CRP, CDAJ/SDAI, SJC (28) and TJC (28) and other parameters of composite scores | approximately 1 year
Quality of life: HAQ-DI score | approximately 1 year
Safety of biologics used in monotherapy: Incidence of adverse events | approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Belgium (14):
  - Aalst
  - Brussels
  - Edegem
  - Genk
  - Ghent
  - Haine-Saint-Paul
  - Kortrijk
  - Liège
  - Merksem
  - Mons
  - Seraing
  - Turnhout
  - Verviers
  - Westmalle